CLINICAL TRIAL: NCT01473979
Title: Delayed Primary Versus Late Secondary Wound Closure in the Treatment of Postsurgical Sternum Osteomyelitis
Brief Title: Delayed Primary Versus Late Secondary Wound Closure in Sternum Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Denis Berdajs, MD, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SternumStudy-CHUV-CCV-1
Record Dates: First submitted 2011-07-11; First posted 2011-11-17 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Mediastinitis
Keywords: cardiac surgery; poststernotomy wound infections; delayed secondary closure of sternum
MeSH Terms: conditions — Mediastinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A) Secondary closure with the vacuum-assisted system (VAC (Active Comparator): after the diagnosis of the poststernotomy wound infection is established the clinical procedure is obtained as follows: firstly the empiric antibiotic therapy with vancomycin is induced. The lab samples including bacteriology test are obtained. Surgical debridement is made until occurrence of tissue bleeding. Finally VAC sponge is implanted wit the negative suction pressure of 75 mmHg.
  The patients are obtained 5 to 7 times to the surgical procedures in time intervals of 48/72 hours. Subsequently when the last three bacteriology samples are negative a delayed primary closure or rectus abdominal muscle flap may be done.
  Interventions: Procedure: Surgical closure of the poststernotomy wound infection
- Arm B) Surgical procedure by delayed primary closure (Active Comparator): In the first step, after the diagnosis of the infection was done, and the empiric antibiotic therapy is induced with vancomycin in the first surgical intervention the sternal wires will be removed, the mediastinum is explored and extensive surgical debridement is performed until occurrence of tissue bleeding.The patients will receive treatment delivered through the VAC system in the first 48 hours following the first surgical intervention, subsequently the wound is closed.
  Interventions: Procedure: Surgical closure of the poststernotomy wound infection

INTERVENTIONS:
Procedure: Surgical closure of the poststernotomy wound infection — Arm A) Secondary closure with the vacuum-assisted system (VAC); The initial surgical revision is done within 24 hours. The first revision with second look and debridement is usually made in 72 hours Subsequently in the following days the wound is stepwise revised during VAC changes.The patients are obtained 5 to 7 times to the surgical procedures in time intervals of 72 hours. Subsequently when the last three bacteriology samples are negative a delayed primary closure or rectus abdominal muscle flap may be done.
  Arm B) Surgical procedure by delayed primary closure; The patients will receive treatment delivered through the VAC system in the first 48 hours following the first surgical intervention, subsequently the wound is closed. after the sternum is closed by using metallic wires, pectoral muscle on both chest parts is mobilized and closed directly over the bone.

SUMMARY:
Sternal osteomyelitis and poststernotomy mediastinitis is a severe and life-treating complication after the cardiac surgery. The incidence of sternal osteomyelitis ranges from 1% to 3% with a high mortality rate from 19% to 29% .

The most devastating complication of the open sternum is the laceration of the right ventricle which has a very high mortality. Additionally destabilizations of the thoracic cage, prolonged immobilization, or substantial surgical trauma are further complications of the conventional strategy (4). In addition, postoperative infections after sternotomy are associated with prolonged hospital stay, increased healthcare costs and impaired quality of patient life, representing an economic and social burden. The emergence of increasing antimicrobial resistant bacteria augments the importance of postsurgical infections since the antimicrobial choices are becoming limited. Furthermore, the incidence of infection is an indicator for the quality of patient care in the international benchmark studies.

Although several therapy strategies are nowadays present in clinical practice, there is a lack of evidence based surgical consensus for treatment of this surgical complication. In most case the poststernotomy mediastinitis is involving surgical revision with debridement, open dressing and/or vacuum assisted therapy. After the granulation tissue on open chest wound was achieved secondary closure and/or reconstruction with vascularized soft tissue flaps such as omentum or pectoral muscle is performed.

It seems there is a need for more effective surgical treatment of poststernotomy wound infections, which may address the prolonged hospitalization and reduce number of surgical interventions and with this also perioperative morbidity. In light of this we propose a randomized study comparing new delay primary closure of the sternum to the secondary vacuum assisted closure.

DETAILED DESCRIPTION:
1. Background

   1.1. Problem of surgical site infection after sternotomy Sternal osteomyelitis and poststernotomy mediastinitis is a severe and life-treating complication after the cardiac surgery. The incidence of sternal osteomyelitis ranges from 1% to 3% (1, 2) with a high mortality rate from 19% to 29% (1, 3).

   The most devastating complication of the open sternum is the laceration of the right ventricle which has a very high mortality. Additionally destabilizations of the thoracic cage, prolonged immobilization, or substantial surgical trauma are further complications of the conventional strategy (4). In addition, postoperative infections after sternotomy are associated with prolonged hospital stay, increased healthcare costs and impaired quality of patient life, representing an economic and social burden. The emergence of increasing antimicrobial resistant bacteria augments the importance of postsurgical infections since the antimicrobial choices are becoming limited. Furthermore, the incidence of infection is an indicator for the quality of patient care in the international benchmark studies.

   Although several therapy strategies are nowadays there is a lack of evidence based surgical consensus for treatment of this surgical complication. In most case the poststernotomy mediastinitis is involving surgical revision with debridement, open dressing, vacuum assisted therapy or closed irrigation. After the granulation tissue on open chest wound was achieved secondary closure and/or reconstruction with vascularized soft tissue flaps such as omentum or pectoral muscle is performed. Both open therapy and the flap implantations may be used as a single-line therapy or as a combination of procedures.

   1.2. Etiology of poststernotomy infections Many mechanisms have been proposed to explain the development of sternal wound infection. These theories include inadequate sternal fixation leading to instability and dehiscence of the overlying skin incision and inadequate surgical drainage. Further theories suggest a localized ischemic osteomyelitis. This theory suggests that sternal wires become loose, leading to sternal instability, which ultimately leads to skin dehiscence and osteomyelitic infection. The most commonly cultured organism is Staphylococcus Aureus.

   Several retrospective and prospective studies have identified factors relating to increasing risk of sternal dehiscence. Patient risk factors include obesity, diabetes mellitus, chronic obstructive lung disease (COPD), chronic cough from tobacco abuse, steroid therapy, hypertension, immunosuppression, and advanced age. Operative risk factors include single or bilateral internal mammary artery (IMA) harvesting (significantly decreases blood supply to ipsilateral hemithorax), prolonged operation, excessive hemorrhage, reoperation, break in sterile technique, and the use of an intra-aortic balloon pump.
2. Objectives

2.1. Study hypothesis The optimal treatment of sternum osteomyelitis has not yet been defined. The aim of this randomized study is to compare the treatment outcome of the delayed primary closure with short-term VAC-therapy (48-72 h) with the late secondary closure with long-term VAC therapy (>14 days).

We hypothesize that the delayed primary closure will have a better outcome than late secondary closure regarding parameters:

* Cure rate (>80% versus <60%)
* Length of hospitalization (≤6 weeks versus >6 weeks)
* Number of surgical interventions (≤4 versus >5)
* In-hospital mortality (5 versus 15%) This combined surgical and active approach has an economic advantage compared to the conventional therapy.

2.2. Aims Primary

1. To compare the treatment outcome (hospital stay, morbidity, mortality and surgical stress load) of the delayed primary closure approach with the late secondary closure Secondary
2. To evaluate side effects of both treatment approaches, and treatment expenses.
3. Study population

   3.1. Ethical aspects The permission from the local Ethical Committee will be obtained before beginning the study. This study will be also registered with www.ClinicalTrials.gov. Patients will be enrolled before randomization 1:1 into each study arm; in each group we will randomly include 40 patients. The randomization is not blind and will be performed by one of the principal investigators. In absence of the principal investigators this may be performed by co-investigators. Surgical procedures in both arms should be standardized. In this way is essential that all the interventions will be performed by main investigator and the co-investigator.

   Arm A) In this group the patients will be treated with the standard surgical treatment. In details the procedure is described under 4.4.

   Arm B) I s the group the patients are treated according to the new concept of the delayed primary sternal closure. The procedure id described under 4.5.
4. Procedures and methods 4.1. Definition of the sternal infection Median sternotomy wound complications vary from sterile wound dehiscence to suppurative mediastinitis. Sternal bone infection, mediastinitis, wound complication, and wound infection have been used synonymously to denote deep sternal wound infection. For the sake of consistency in comparing data from various reports, definitions of sternal wound complications are as follows (8,9,10).

Ad 1) Mediastinal dehiscence: median sternotomy wound breakdown in the absence of clinical or microbiologic evidence of infection.

Ad 2) Mediastinal wound infection: clinical or microbiologic evidence of infected presternal tissue and sternal osteomyelitis, with or without mediastinal sepsis and with or without unstable sternum. Subtypes include:

A) superficial wound infection: wound infection confined to the subcutaneous tissue B) deep wound infection (mediastinitis): wound infection associated with sternal osteomyelitis with or without infected retrosternal space. Deep sternal wound infections, or mediastinitis, is classified into four subtypes based on the time of first presentation, the presence or absence of risk factors, and whether previous attempts at treating the condition have failed (Table 1).

Sternal wound infection will be considered:

The definition of mediastinitis has been established by the Center for Disease Control and Prevention in the USA (11). According to these guidelines, diagnosis of mediastinitis requires at least one of the following:

Ad 1) an organism isolated from culture of mediastinal tissue or fluid; Ad 2) evidence of mediastinitis seen during operation; Ad 3) one of the following conditions: chest pain, sternal instability, or fever (>38 8C), in combination with either purulent discharge from the mediastinum or an organism isolated from blood culture or culture of mediastinal drainage.

4.2. Outline of the surgical procedures Patients with suspected sternal osteomyelitis will be hospitalized and the following diagnostic procedures will be performed: laboratory blood tests (leukocytes, CRP, creatinin, AST, ALT, CK), computed tomography (CT) of the sternum, wound swab.

After the diagnosis is secured the patients will receive an information consent form of the study. Subsequently they will be randomly included in one of the surgical arms.

4.3. Current treatment strategy of poststernotomy infections During the past years, vacuum-assisted closure (VAC) wound therapy has emerged as a treatment for open septic wounds. It is a non-invasive system that helps promote wound healing by delivering negative pressure the application of this subatmospheric form of treatment has, several advantageous as compared to the conventional treatment. VAC therapy allows open drainage that continuously absorbs exudate with simultaneous stabilization of the chest and isolation of the wound. This therapy induces the building of the granulation tissue which in majority is a result of the reduced oedema and increased blood flow in the adjacent tissue. Furthermore, VAC therapy approximates the wound edges and provides a mass filling effect with a low degree of surgical trauma, without establishing a new wound (e.g., abdominal wound in omental flaps) (5,6). In the recent literature the mean hospitalization of the patients being treated with the VAC therapy was 25 ± 20 days with overall mortality of 15%.

4.4. Arm A) Secondary closure with the vacuum-assisted system (VAC) Nowadays after the diagnosis of the poststernotomy wound infection is established the clinical procedure is obtained as follows: firstly the empiric antibiotic therapy with vancomycin is induced. The lab samples including bacteriology test are obtained. The initial surgical revision is done within 24 hours. Intraoperatively from the surgical field again tissue samples are sent for bacteriology investigation to determine the antibiotic pattern resistance. All sternal wires are removed. Surgical debridement is made until occurrence of tissue bleeding. Careful and extensive cleaning of the wound is performed using saline solution at 37°C degrees Celsius and the solution of 50% betadine and saline solution (1:1 Betadine:H20). Finally VAC sponge is implanted with negative suction pressure of 75 mmHg. Postoperatively chest X-ray is obtained, in the first 24 hours the lab samples with CRP and whit blood cell count is performed. The first revision with second look and debridement is usually made in 48 hours. Subsequently in the following days the wound is stepwise revised during VAC changes (every 48/72 hours) a sharp spoon and necrotic bone is removed when necessary, but extensive sternectomy is avoided. At each revision tissue samples are obtained for microbiological investigations.

According to the patients general situation they are extubated immediately after VAC therapy initiation and are staying on the intensive care unit for about 24 hours. The patients are obtained 5 to 7 times to the surgical procedures in time intervals of 48/72 hours. Subsequently when the last three bacteriology samples are negative a delayed primary closure by usage of Kryptonite biocompatible adhesive glue (Doctors Research Group Inc, Southbury, CT)- if needed for sternal stabilization- or rectus abdominal muscle flap may be done. As far the antibiogram is known, the specific antibiotic therapy is induced.

4.5. Arm B) Surgical procedure by delayed primary closure As compared to the previous therapy modalities mentioned under 2.2 and 1.3 the new method has an advantage of the surgical wound healing by delayed primary intention.

In the first step, after the diagnosis of the infection was done, and the empiric antibiotic therapy is induced with vancomycin in the first surgical intervention the sternal wires will be removed, the mediastinum is explored and extensive surgical debridement is performed until occurrence of tissue bleeding. Careful and extensive cleaning of the wound was performed using saline solution at 37°C degrees Celsius and the solution of 50% betadine and saline solution (1:1 Betadine:H20), at least 3 samples (tissue biopsies) are taken for microbiology. The patients will receive treatment delivered through the VAC system in the first 48 hours following the first surgical intervention. Subsequently the wound is closed.

We begin with dissection and elevation of the pectoralis major muscle and corresponding subcutaneous flap through diathermy. Dissection is performed from the median line along the costal grid, up to two thirds of the anterior chest wall, preserving the humeral insertion, thoracoacromial vascular bundle and pectoralis minor muscle. Note at this area are very important vascular connections areas between the internal thoracic artery, acromial artery and the lateral thoracic artery which should be preserved. At inferior plane, the pectoralis major muscle will be raised - including the anterior rectus fascia - and down up to the xiphoid process. The upper segment of the anterior rectum will be raised with the pectoralis major muscle. The intercostal perforating arterial branches will be preserved also. A silicon drain tube is placed in the retrosternal space if this is possible. In patients with fracture or asymmetry of the sternum incision, osteosynthesis is performed using the "Robiscek" technique. Then two suction drains were placed below the muscular plane upon the costal grid for drainage of the large area of detachment of the musculoaponeurotic layer The suture of the pectoral fascia should be tension free, continuous suture with resorbable material (Vicryl 3-0). The subcutaneous tissue is closed over the drainage, with separate subcutaneous suture. The skin is closed with non-resorbable suture analog to the "Allgöver" suture. These sutures are removed between the 12 and 14 postoperative days.

Thus the results of the bacteriology are known in most cases after the first 48 hours the specific antibiotic therapy, according to the results of the bacteriology results may be introduced.

4.6 General considerations

Contraindication for closure of the chest:

Wounds with active purulence require extensive debridement prior to flap coverage and/or rigid fixation. Additional contraindications for sternal reconstruction are found in patients who are unstable for surgery, including those with poor pulmonary function, poor cardiac reserve, or terminal illness. Hemodynamic stability is required for surgical intervention in patients with sternal dehiscence.

4.7. Early perioperative management in the 48 hours

Transfer to the ICU:

After each definitive sternal closure the patients will be transferred to the ICU for the hemodynamical observation in the first 24 hours. Beside the followings are considered as indications to transfer on ICU.:

Preoperative sepsis, intraoperative hemodynamical instability or/and need for catecholamines, intraoperative need for massive transfusion, rupture of the ventricular cavities (left or right), need for emergency cardiopulmonary bypass.

Transfer to the intermediate car Hemodynamical and pulmonary stable patients will be extubated in the operating room, and will be transferred to the intermediate care unit of the department of cardiovascular surgery.

General considerations Independently in both investigation groups Arm A) and Arm B) postoperatively X-ray of the thorax will be obtained after the transfer. In the first 24 hours, the lab samples will be obtained (CRP, anticoagulation, white blood cell cont, hemoglobin, hematocrit, ASAT, ALAT, yGT, Creatinine, Urea, and anticoagulation tests PTT, TP). Respiratory physiotherapy will be obtained 24 hours after the surgical revision.

Open chest patients should not be mobilized out of the bed, however the chest elevation and mobilization of 45 to 90° is aloud.

After definitive closure of the chest the patient may be fully mobilized after the first 48 hours, or after the transfer to the ward.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or more
* Who has been operated on the open heart and received a total or partial median sternotomy
* Informed consent has been obtained, subject is willing to follow protocol study treatment regimen, and comply with all planned follow-up assessments
* Not self-determined patients are not exclusion criteria

Exclusion Criteria:

* after heart transplantation or other orthotropic transplantation procedure
* superficial wound infections (see definition at 4.1)
* Sterile open wound dehiscence's without any sign of local or systematic infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
In hospital Mortality | 30 days

SECONDARY OUTCOMES:
in hospital stay | 30 days
number of surgical interventions during hospitalization | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Cardiovascular Surgery, University Hospital Lausanne (CHUV), Lausanne, Switzerland